CLINICAL TRIAL: NCT04445038
Title: A Randomized, Double-blind, Placebo-controlled Parallel Trial of Safety, Tolerability and Pharmacokinetic of Recombinant Anti-IL-5 Humanized Monoclonal Antibody by Single Subcutaneous Injection in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic of Recombinant Anti-IL-5 Humanized Monoclonal Antibody Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-610-HH-I-01
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-06

CONDITIONS: add-on Maintenance Treatment of Patients With Severe Eosinophilic Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 610 group (Experimental): Participants will be administered with 0.03mg/kg, 0.2mg/kg, 1.0mg/kg, 3.0mg/kg, 5.0mg/kg, 7.5mg/kg of 610 by subcutaneous injection. Subjects will be followed for 84 days.
  Interventions: Drug: 610
- controll group (Placebo Comparator): Participants will be administered with 0.2mg/kg, 1.0mg/kg, 3.0mg/kg, 5.0mg/kg, 7.5mg/kg placebo once by subcutaneous injection. Subjects will be followed for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 610 — Recombinant anti-IL-5 Humanized Monoclonal Antibody
  Arms: 610 group
Drug: Placebo — Placebo
  Arms: controll group

SUMMARY:
This study is Safety, Tolerability and Pharmacokinetic of Recombinant anti-IL-5 Humanized Monoclonal Antibody injection in Healthy Subjects. There are 6 Groups as follows: 0.03mg/kg (S1), 0.2mg/kg (S2), 1.0mg/kg (S3), 3.0mg/kg (S4), 5.0mg/kg (S5) and 7.5mg/kg (S6); and 2 subjects were included in the S1 group (both received study drugs); 10 subjects were included in each of the S2 ~ S6 groups (of which 8 received study drugs and 2 received placebo). Pharmacokinetics and Anti-drug antibody (ADA) data will be collected; Drug safety, tolerance, efficacy and immunogenicity for healthy subjects will be evaluated.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled parallel trial of safety, tolerability and pharmacokinetic of Recombinant anti-IL-5 Humanized Monoclonal Antibody by single subcutaneous injection with six different doses in healthy subjects. There are 6 groups as follows: 0.03mg/kg (S1), 0.2mg/kg (S2), 1.0mg/kg (S3), 3.0mg/kg (S4), 5.0mg/kg (S5) and 7.5mg/kg (S6); and 2 subjects were included in the S1 group (both received study drugs); 10 subjects were included in each of the S2 ~ S6 groups (of which 8 received study drugs and 2 received placebo). In each group, two subjects were sentinels (1 received the study drug and 1 placebo). Pharmacokinetics and Anti-drug antibody (ADA) data will be collected; Drug safety, tolerance, efficacy and immunogenicity for healthy subjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy participants, male or female, aged 18 to 55 (including both ends)
* The body mass index (BMI) is in the range of 19.0~28.0 kg•m-2 (including both ends), and the weight of men is generally not less than 50kg, while the women is generally not less than 45kg
* Male participants and their partners or female participants must agree to take one or more non-drug contraceptives (such as complete abstinence, contraceptive rings, partner ligation, etc.) , and there is no sperm donation or egg donation plan
* Participants should fully understand the purpose, nature, methods and possible adverse reactions of the trial, volunteer to participate in the trial and sign the informed consent
* Participants could communicate well with the researchers and compliance with the trial

Exclusion Criteria:

* Those who are allergic to the study drug and any of its excipients. Subjects who have a history of allergy to monoclonal antibodies, and with allergies (multiple drugs and food allergies)
* Subjects who have or are currently suffering from any serious clinical diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities or any other that can interfere with the study results
* Those who have undergone surgery within the 3 months prior to the trial that will affect the absorption, distribution, metabolism, and excretion of the drug; or those who have undergone surgery within 4 weeks prior to the trial, or plan to undergo surgery during the study
* Positive for Hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HbcAb), anti- Hepatitis C virus antibodies (HCV), or anti-human immunodeficiency virus (HIV)
* Alcoholics or frequent drinkers within 6 months before the trial, drinking more than 14 units per week (1 unit alcohol ≈360 mL beer or 45 mL spirits with 40% alcohol content or 150 mL wine), or couldn't prohibit alcohol during the trial or alcohol breath test results greater than 0.0 mg / 100 mL
* Those who smoked more than 5 cigarettes per day during the 3 months before screening, or who cannot stop using any tobacco products during the trial
* Drug abusers or those who have used soft drugs (such as marijuana) within 3 months or took hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the trial, or have positive drug abuse screening (morphine, methamphetamine , Ketamine, ecstasy, marijuana)
* Has taken any prescription medicine, non-prescription medicine, Chinese herbal medicine or health products (vitamins, cod liver oil, etc.) within 14 days before administration
* Has received any monoclonal antibody drugs within 5 half-lives before administration
* Has a history of vaccination within 4 weeks before dosing, or intend to receive vaccines during the study
* Has parasitic infection at present and within 3 months before dosing
* Was previously enrolled in other clinical trials within 3 months
* Blood donors or subjects who lost a lot of blood (> 400 mL, except for women's physiological period) or those who received blood transfusion or used blood products within 3 months
* Can't tolerate venipuncture or has a history of halo needles and halo blood
* Has known or suspected pregnancy or lactation
* Abnormal vital signs (SBP <90 mmHg or ≥140 mmHg, DBP <55 mmHg or ≥90 mmHg; heart rate <50 bpm or> 100 bpm; body temperature (ear temperature) <35.4℃ or > 37.7℃) or abnormal ECG (QTcB male ≥450 ms, female ≥460 ms) or physical examination, laboratory examination, and abdominal ultrasound examination are clinically significant (according to the judgment of clinical research doctors)
* Subjects who are unsuited to the study for any reason, judged by the investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to 84 days
  Maximum Plasma Concentration of 610
Tmax | up to 84 days
  Time to Maximum Plasma Concentration of 610
AUC | up to 84 days
  Area Under the Curve of 610
t1/2 | up to 84 days
  Half life of 610 in blood
CL/F | up to 84 days
  Plasma clearance of 610
Vd/F | up to 84 days
  Apparent Volume of Distribution of 610
AE | up to 84 days
  To monitor adverse events (AEs) per the NCI CTCAE 5.0.

SECONDARY OUTCOMES:
Immunogenicity | up to 84 days
  Percentage of ADA positive and determination of ADA titer as well as Nab
EOS | up to 84 days
  Compare the changes of EOS levels with the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Ding, D.M., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided